CLINICAL TRIAL: NCT05269784
Title: Minimally Invasive Lung Surgery Under ERAS With Completely Tubeless Protocol Compared With That With Partially Tubeless Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Completely Tubeless ZYP
Record Dates: First submitted 2022-02-26; First posted 2022-03-08 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-02

CONDITIONS: Lung Diseases; ERAS; Surgery
Keywords: tubeless; enhanced recovery after surgery (ERAS); lung surgery; no intubation; urinary catheter
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Completely Tubeless Group (Experimental): minimally invasive lung surgery under ERAS with completely tubeless protocol: no intubation, no urinary catheter, move the chest drainage as fast as possible according the ERAS guideline on the premise of safety.
  Interventions: Procedure: Minimally Invasive Lung Surgery Under ERAS With Completely Tubeless Protocol
- Partially Tubeless Group (Active Comparator): minimally invasive lung surgery under ERAS with partially tubeless protocol.
  Interventions: Procedure: Minimally Invasive Lung Surgery Under ERAS With partially Tubeless Protocol

INTERVENTIONS:
Procedure: Minimally Invasive Lung Surgery Under ERAS With Completely Tubeless Protocol — Minimally Invasive Lung Surgery Under ERAS With Completely Tubeless Protocol
  Arms: Completely Tubeless Group
Procedure: Minimally Invasive Lung Surgery Under ERAS With partially Tubeless Protocol — Minimally Invasive Lung Surgery Under ERAS With partially Tubeless Protocol
  Arms: Partially Tubeless Group

SUMMARY:
Previous studies have shown the feasibility of ERAS on minimally invasive lung surgery, but it is unknown whether completely tubeless protocol is safe and better. This study aimed to determine whether completely tubeless protocol is feasible and beneficial for minimally invasive lung surgery, compared with partially tubeless protocol.

ELIGIBILITY:
Inclusion Criteria:

(I) Wedge resection or sub-lobar resection or lobectomy is considered as the primary surgical strategy. The operation ideally should not exceed 2 hours; (II) No absolute age limit; (III) Patients with Eastern Cooperative Oncology Group (ECOG) physical performance score of ≤2 points; (IV) P a t i e n t s w i t h a n A m e r i c a n S o c i e t y o f Anesthesiologists Standard (ASA) grade of ≤ III; (V) Body mass index (BMI) <30 kg/m2; (VI) Patients with no clinically significant cardiac history, such as ischaemic heart disease, valvular heart disease, rhythm disturbances such as frequent atrial fibrillation or premature ventricular contractions (PVCs). Patients with significant cardiac history should be optimized according the relevant guidelines before surgery is considered; (VII) Normal cardiopulmonary function [predicted forced expiratory volume in the first second (FEV1%) >50% and ejection fraction (EF) >50% of predicted value]. Resting blood gas analysis showing arterial partial pressure of oxygen (PaO2)≥75 mmHg and arterial partial pressure of carbon dioxide (PaCO2) <45 mmHg; (VIII) Normal renal function and no history of urological problems.

Exclusion Criteria:

(I) Patient-related factors: (i) Patients who refuse surgery and/or the anesthesia protocols; (ii) Coagulopathy, hypoxemia (PaO2 <60 mmHg), hypercapnia [arterial carbon dioxide tension (PaCO2) >50 mmHg], or elevated risk of regurgitation (<6 hours of fasting) preoperatively or combined with gastroesophageal reflux disease; neurological disorders; (iii) Severe acute pulmonary infection or tuberculosis; (iv) Relative contraindications: upper airway secretions or persistent cough, spinal deformity, or brain edema (if thoracic epidural anesthesia is to be used); (v) History of ipsilateral surgery and other conditions which can result in extensive pleural adhesion; (vi) Phrenic nerve paralysis on the non-operated side should be viewed as a contraindication to VATS; (vii) History of urological conditions increasing the need for urinary catheterization; (viii) Significant cardiac history. (II) Anesthesia-related factors: (i) Allergy to local anesthesia; (ii) Any contraindication to the regional anesthesia.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
urinary irritation and urinary tract infection | within a week after surgery
  incidence rate
0-degree discomfort | within 3 days after surgery
  proportion
duration of postoperative hospital stay | within 7 days after surgery
  days
pneumonia | within 7 days after surgery
  incidence rate
operation time | within 150 minutes
  minutes
bleeding volume | during surgery
  ml ml
volume of drainage | within 7 days after surgery
  ml
Pain degree | within 7 days after surgery
  On a scale of 1 to 10
drainage duration time | within 7 days after surgery
  days

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Shandong University, Jinan, Shandong, China

REFERENCES:
- [Derived] Zhao Y, Shan L, Zhang W, Li P, Li N, Zhang H, Peng C, Cong B, Zhao X. Minimally invasive lung surgery with an intraoperative completely or partially tubeless protocol: randomized clinical trial. BJS Open. 2024 Dec 30;9(1):zrae132. doi: 10.1093/bjsopen/zrae132. PMID 39924850